CLINICAL TRIAL: NCT02221375
Title: Safety, Tolerability and Pharmacokinetics of Multiple Rising Inhalative Doses of Butylated Hydroxytoluene Via Respimat Soft MistTM Inhaler B (Sub-study 1) and Safety, Tolerability and Pharmacokinetics of Multiple Rising Inhalative Doses of BI 54903 XX Via Respimat Soft MistTM Inhaler B as Randomised, Double-blind, Placebo-controlled Phase I Trial in Healthy Male Volunteers (Main Study) and Comparison of Systemic Exposure Following a Single Dose of BI 54903 XX Via Respimat Soft MistTM Inhaler B and of a Single Dose of Ciclesonide Via MDI (Randomised, Open-label, Two-way Crossover Sub-study 2)
Brief Title: Safety, Tolerability and Pharmacokinetics of Multiple Rising Doses of Butylated Hydroxytoluene and BI 54903 XX Via Respimat® Soft MistTM Inhaler B in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1256.1
Record Dates: First submitted 2014-08-19; First posted 2014-08-20 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
MeSH Terms: interventions — ciclesonide

ARMS (9):
- BHT low (Experimental)
  Interventions: Drug: BHT low
- BHT medium (Experimental)
  Interventions: Drug: BHT medium
- BHT high (Experimental)
  Interventions: Drug: BHT high
- BI 54903 XX low (Experimental)
  Interventions: Drug: BI 54903 XX low
- BI 54903 XX medium 1 (Experimental)
  Interventions: Drug: BI 54903 XX medium 1
- BI 54903 XX medium 2 (Experimental)
  Interventions: Drug: BI 54903 XX medium 2
- BI 54903 XX high (Experimental)
  Interventions: Drug: BI 54903 XX high
- BI 54903 XX medium single dose (Experimental)
  Interventions: Drug: BI 54903 XX medium 2
- Ciclesonide (Active Comparator)
  Interventions: Drug: Ciclesonide

INTERVENTIONS:
Drug: BHT low
  Arms: BHT low
Drug: BHT medium
  Arms: BHT medium
Drug: BHT high
  Arms: BHT high
Drug: BI 54903 XX low
  Arms: BI 54903 XX low
Drug: BI 54903 XX medium 1
  Arms: BI 54903 XX medium 1
Drug: BI 54903 XX medium 2
  Arms: BI 54903 XX medium 2; BI 54903 XX medium single dose
Drug: BI 54903 XX high
  Arms: BI 54903 XX high
Drug: Ciclesonide
  Arms: Ciclesonide

SUMMARY:
The objective of the study was to investigate safety, tolerability and pharmacokinetics of butylated hydroxytoluene (BHT) (sub-study 1) administered via Respimat® Soft MistTM Inhaler B (SMI B); to assess safety, tolerability and pharmacokinetics of multiple rising doses of BI 54903 XX administered via Respimat® SMI B (main study), and to compare systemic exposure of single dose BI 54903 XX administered via Respimat® SMI B (sub-study 2) with single dose Alvesco® (ciclesonide) administered via HFA-134a propellant metered dose inhaler (MDI).

ELIGIBILITY:
Inclusion Criteria:

* Healthy males based upon a complete medical history, including the physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead Electrocardiogram (ECG) and clinical laboratory tests
* Age >= 21 and <= 50 years
* BMI >= 18.5 and <= 29.9 kg/m2
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (>24 h) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of drugs that could reasonably influence the results of the trial within 10 days prior to administration or during the trial (based on the knowledge at the time of protocol preparation)
* Participation in another trial with an investigational drug within 2 months prior to administration or during the trial
* Smoker (>10 cigarettes or >3 cigars or >3 pipes per day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (more than 60 g per day)
* Drug abuse
* Blood donation (>100 mL within 4 weeks prior to administration or during the trial)
* Excessive physical activities (within 1 week prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of the trial site
* Bacterial and viral infections of the lung, including active or latent tuberculosis

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2008-06; Primary Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events | up to 21 days after last drug administration
Number of patients with clinically significant findings in vitals signs | up to 21 days after last drug administration
Number of patients with clinically significant findings in ECG | up to 21 days after last drug administration
Number of patients with clinically significant findings in laboratory tests | up to 21 days after last drug administration
Investigator assessed tolerability on a 4-point scale | up to 21 days after last drug administration
Change in airway resistance (Raw) | baseline, after 80 hours

SECONDARY OUTCOMES:
Cmax (maximum measured concentration in plasma) | up to 24 hours after last drug administration
tmax (time from dosing to maximum measured concentration in plasma) | up to 24 hours after last drug administration
AUCτ (area under the concentration-time curve in plasma over a uniform dosing interval τ) | up to 24 hours after last drug administration
AUC0-inf (area under the concentration-time curve in plasma over the time interval from 0 extrapolated to infinity) | up to 24 hours after last drug administration
AUCt1-t2 (area under the concentration-time curve in plasma over the time interval from time t1 to time t2) | up to 24 hours after last drug administration
AUC0-tz (area under the concentration-time curve in plasma over the time interval from 0 to the last quantifiable concentration at tz) | up to 24 hours after last drug administration
%AUCtz-∞ (the percentage of the AUC 0-∞ that is obtained by extrapolation) | up to 24 hours after last drug administration
λz (terminal rate constant in plasma) | up to 24 hours after last drug administration
t1/2 (terminal half-life in plasma) | up to 24 hours after last drug administration
MRTih (mean residence time in the body after inhalation administration) | up to 24 hours after last drug administration
CL/F (apparent clearance in plasma following inhalation administration) | up to 24 hours after last drug administration
Vz/F (apparent volume of distribution during the terminal phase λz following inhalation administration) | up to 24 hours after last drug administration
Aet1-t2 (amount that is eliminated in urine from the time point t1 to time point t2) | up to 24 hours after last drug administration
fet1-t2 (fraction that is eliminated in urine from time point t1 to time point t2) | up to 24 hours after last drug administration
CLR,t1-t2 (renal clearance from the time point t1 until the time point t2) | up to 24 hours after last drug administration
Accumulation ratio based on Cmax (RA,Cmax) | up to 24 hours after last drug administration
Accumulation ratio based on AUC (RA,AUC) | up to 24 hours after last drug administration
Linearity index (LI) | up to 24 hours after last drug administration
Metabolite-to-parent ratio for Cmax (RCmax,Met) | up to 24 hours after last drug administration
Metabolite-to-parent ratio for AUC (AUCt1-t2,Met) | up to 24 hours after last drug administration